CLINICAL TRIAL: NCT00517075
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Negative Symptoms and Social Dysfunction in Schizophrenia Patients
Brief Title: Treatment of Negative Symptoms of Schizophrenia With Transcranial Magnetic Stimulation (TMS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to adequately recruit subjects.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5977R
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Transcranial Magnetic Stimulation; Repetitive Transcranial Magnetic Stimulation; Schizophrenia; Schizoaffective Disorder; Treatment; Negative Symptoms; Social Dysfunction; TMS; rTMS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): high frequency rTMS to the left infero-parietal lobe, active/sham condition randomized (2:1), double-blind
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- B (Active Comparator): Active high frequency rTMS to the left dorsolateral prefrontal cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- C (Sham Comparator): Sham (placebo) high frequency rTMS to the left dorsolateral prefrontal cortex or left infero-parietal lobe, active/sham condition randomized (2:1), double-blind
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Open cross over high frequency rTMS (Experimental): Following the randomization phase with three arms, subjects who did not respond, have the possibility of receiving open active treatment to the target that they did not receive treatment to in the randomization phase. (i.e. randomized to IPL --> open phase DLPFC and vice versa)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
  Other Names: Magstim Rapid 2
  Arms: A
Device: Transcranial Magnetic Stimulation (TMS) — For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
  Other Names: Magstim Rapid 2
  Arms: B
Device: Transcranial Magnetic Stimulation (TMS) — For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
  Other Names: Magstim Rapid 2
  Arms: C
Device: repetitive transcranial magnetic stimulation — For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
  Other Names: MagStim Rapid2
  Arms: Open cross over high frequency rTMS

SUMMARY:
This study will test whether repetitive transcranial magnetic stimulation (rTMS) is helpful in treating negative symptoms and social deficits of schizophrenia. This will be the first rTMS study to assess social function and social cognition.

1. Hypoactivity in the dorsolateral prefrontal cortex (DLPFC) has been implicated in generating the negative symptoms of schizophrenia. Abnormalities in the left inferior parietal lobe (IPL) have also been associated with negative symptoms. We hypothesize that high frequency rTMS applied to the hypoactive left DLPFC or to the left IPL in individuals with schizophrenia will reduce negative symptom severity more than sham (placebo) rTMS as assessed by the Positive and Negative Syndrome Scale (PANSS) negative symptoms subscale.
2. We hypothesize that high frequency rTMS applied to the left DLPFC or to the left IPL in schizophrenia patients will improve social dysfunction more than sham (placebo) rTMS as assessed by the Social Adjustment Scale, the Social Adaptation Self-Evaluation Scale and the Social Functioning Scale.

DETAILED DESCRIPTION:
Most treatments for schizophrenia are helpful in treating positive symptoms (e.g. hallucinations), whereas negative symptoms (e.g. low social drive) are only partially responsive to medication. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive way of stimulating the brain that has been FDA approved for the treatment of depression and has shown promise in schizophrenia.

In rTMS therapy, a device called a "magnetic stimulator" provides electrical energy to a magnetic coil that delivers a magnetic field. When the coil is placed against the surface of the head, the magnetic field can cause parts of the brain to either increase or decrease in activity, depending on how quickly the magnetic pulses are delivered. This study is designed to test whether high-frequency rTMS delivered to an area near the front of the head, called the dorsolateral prefrontal cortex, can improve the "negative symptoms" of schizophrenia, which include decreased thinking, difficulty motivating, and social withdrawal.

Participation in the first phase of the study consists of sessions lasting about 45 minutes per day, 5 days a week, for 4 weeks. Twenty-four subjects will be randomly assigned to receive four weeks of either active (real) rTMS or inactive (sham) rTMS. Patients will receive magnetic resonance imaging (MRI) of their brains to help locate where the rTMS should be applied. Symptoms will be rated at baseline, during the rTMS course, and at the end of the 4 weeks. Patients who do not meet response criteria after the four weeks of the randomized phase will be offered active (real) daily rTMS for an additional four weeks in the open phase of the study. All patients will have two monthly repeat assessments after their last rTMS session to examine the persistence of benefit.

We will also collect measures of motor cortex excitability (performed with single pulse TMS) at baseline, at the end of the randomized and, if applicable, the open study phase, and at each of the two follow-up assessments to determine whether changes in these measures correlate with clinical improvement.

In addition, we will look at brain dynamics using electroencephalography (EEG) pre- and post-rTMS in the first and last sessions of each study phase. We will also assess the effects of rTMS on cigarette use, as schizophrenia patients are known to have increased prevalence of nicotine dependence. There is also preliminary evidence that high frequency rTMS to the left DLPFC decreases cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Male or female inpatients or outpatients, 18 to 55 years of age.
* Primary diagnosis by DSM-IV criteria for Schizophrenia or Schizoaffective Disorder.
* Capacity and willingness to give informed consent.
* Engaged in ongoing treatment with a psychiatrist.
* PANSS negative symptoms subscale score of ≥ 15.
* English speaking.
* Patients must have stable symptoms as defined by not requiring a change in antipsychotic medication for at least 4 weeks or at least 2 weeks for other psychotropic agents (e.g. antidepressants) prior to entering the study. Patients will not be included in the study if the research team thinks that modifications could be made to maximize their medication regimen at initial evaluation.
* Able to adhere to the treatment schedule.
* Able to commute to NYC for daily treatments (Monday - Friday) for at least 4 weeks.

Exclusion Criteria:

* Individuals diagnosed by the investigator with the following conditions (current unless otherwise stated): Current affective disorder including Major Depressive Disorder, Bipolar Affective Disorder; substance abuse or dependence within the past year (except nicotine and caffeine).
* An Axis II Personality Disorder, which in the judgment of the investigator may hinder the patient in completing the procedures required by the study protocol.

Other exclusion criteria include those common to every TMS protocol:

* Individuals with a clinically defined neurological disorder or insult including, but not limited to: Any condition likely to be associated with increased intracranial pressure; Space occupying brain lesion; Any history of seizure EXCEPT those therapeutically induced by ECT; History of cerebrovascular accident; Transient ischemic attack within two years; Cerebral aneurysm; Dementia; Parkinson's disease; Huntington's chorea; or Multiple sclerosis.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), history of epilepsy or seizure in first-degree relatives, having metal inside the head, or history of significant head trauma with loss of consciousness for 5 minutes.
* Prior adverse reaction to TMS.
* History of treatment with rTMS therapy for any disorder.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* Current illicit drug use.
* Clinically significant laboratory abnormality, in the opinion of the investigator. (Note: Clinically significant laboratory abnormality refers to patient lab results that fall outside the established normal ranges, may be indicative of the presence of a medical condition, and are not thought to reflect an artifact or routine lab error (e.g. hemolysis). Results of laboratory tests are reviewed by the study physician prior to any treatment. Abnormal lab results of clinical significance that cannot be resolved (e.g. by repeating the test to rule out laboratory error or poor quality of the original sample) will lead to exclusion from the study.)
* Known or suspected pregnancy.
* Women who are breast-feeding.
* Women of child-bearing potential not using a medically accepted form of contraception when engaging in sexual intercourse.
* Wearing medicinal skin patches during the MRI scan.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2004-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arielle D. Stanford, MD, Principal Investigator — New York State Psychiatric Institute / Columbia University College of Physicians and Surgeons
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Hajak G, Marienhagen J, Langguth B, Werner S, Binder H, Eichhammer P. High-frequency repetitive transcranial magnetic stimulation in schizophrenia: a combined treatment and neuroimaging study. Psychol Med. 2004 Oct;34(7):1157-63. doi: 10.1017/s0033291704002338. PMID 15697042
- [Background] Sachdev P, Loo C, Mitchell P, Malhi G. Transcranial magnetic stimulation for the deficit syndrome of schizophrenia: a pilot investigation. Psychiatry Clin Neurosci. 2005 Jun;59(3):354-7. doi: 10.1111/j.1440-1819.2005.01382.x. PMID 15896231
- [Background] Jin Y, Potkin SG, Kemp AS, Huerta ST, Alva G, Thai TM, Carreon D, Bunney WE Jr. Therapeutic effects of individualized alpha frequency transcranial magnetic stimulation (alphaTMS) on the negative symptoms of schizophrenia. Schizophr Bull. 2006 Jul;32(3):556-61. doi: 10.1093/schbul/sbj020. Epub 2005 Oct 27. PMID 16254067
- See also: Division of Brain Stimulation and Therapeutic Modulation, Columbia University — http://www.brainstimulation.columbia.edu/
- See also: Department of Psychiatry, Columbia University — http://columbiapsychiatry.org/
- See also: New York State Psychiatric Institute — http://www.nyspi.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Groups:
- High Frequency rTMS: high frequency rTMS to the left infero-parietal lobe, active/sham condition randomized (2:1), double-blind
  Transcranial Magnetic Stimulation (TMS): For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
- Active High Frequency rTMS: Active high frequency rTMS to the left dorsolateral prefrontal cortex
  Transcranial Magnetic Stimulation (TMS): For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
- Sham/Placebo: Sham (placebo) high frequency rTMS to the left dorsolateral prefrontal cortex or left infero-parietal lobe, active/sham condition randomized (2:1), double-blind
  Transcranial Magnetic Stimulation (TMS): For rTMS, the coil is held flat on the scalp. 40 trains of 10 Hz rTMS will be delivered in trains lasting 4 seconds, with an intertrain interval of 26 seconds, for a total of 20 minutes (1600 pulses per day) at 100% motor threshold. Subjects will receive rTMS once a day, 5 days a week, for 4 weeks. During the first week of rTMS sessions only, in the event that the patient cannot tolerate these stimulation parameters, intensity relative to motor threshold may be titrated downward, in a masked fashion, to 80%, with all other dose parameters remaining the same.
Period: Overall Study
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Continuous
Gender
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement of Negative Symptoms (Positive and Negative Syndrome Scale [PANSS] Negative Symptoms Subscale) Relative to Pre-treatment Baseline.
Time Frame: At baseline, every 2 weeks during rTMS sessions, and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Global Clinical Improvement
Time Frame: At baseline, every 2 weeks during rTMS sessions, and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Social Functioning
Time Frame: At baseline, every 2 weeks during rTMS sessions, and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Depression
Time Frame: At baseline, every 2 weeks during rTMS sessions, and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Theory of Mind
Time Frame: At baseline and the end of each study phase (random and open)
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Smoking Behaviors
Time Frame: At baseline, every 2 weeks during rTMS sessions, and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Cognitive Function
Time Frame: At baseline, the first and last rTMS sessions of each study phase (random and open), and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Cortical Excitability
Time Frame: At baseline, every 2 weeks during rTMS sessions, and at monthly follow-up visits.
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | High Frequency rTMS | Active High Frequency rTMS | Sham/Placebo | Open Cross Over High Frequency rTMS
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes